CLINICAL TRIAL: NCT07351578
Title: Knee Arthroplasty Recovery With Transcranial Direct Current Stimulation: A Randomized Controlled Pilot Trial
Brief Title: Knee Arthroplasty Recovery With Transcranial Direct Current Stimulation
Acronym: KART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: AFP Innovation Fund (Other); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Karim Ladha, MD MSc FRCPC, Women's College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTO 5609
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Knee Arthroplasty; Transcranial Direct Current Stimulation; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, double-blinded, active-placebo controlled trial with two parallel arms.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As noted above, only the company created the randomization will be aware of allocation assignment. The participant, Investigator, surgeon and outcomes assessors will be blinded to minimize bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based tDCS (Experimental): receives active stimulation
  Interventions: Device: Active tDCS Stimulation
- Sham tDCS (Placebo Comparator): receives non-active stimulation
  Interventions: Device: Sham tDCS Stimulation

INTERVENTIONS:
Device: Active tDCS Stimulation — Participants will have electrodes positioned on their scalp at C3, C4 (primary motor cortices) and Oz (occipital cortex) according to the international 10-20 EEG system. They will receive active transcranial direct current stimulation (tDCS) to the primary motor cortex (M1) opposite the surgical site, with the Oz electrode serving as the return. Stimulation will be delivered at 2 mA for 20 minutes, including a 15-second ramp-up at the start and a 15-second ramp-down at the end. The PlatoWork 2.0 tDCS Neurostimulator headset will be used to administer the stimulation.
  Arms: Home-based tDCS
Device: Sham tDCS Stimulation — Participants will receive sham (inactive) transcranial direct current stimulation (tDCS) using the PlatoWork 2.0 tDCS Neurostimulator headset at home. The headset is identical to the active device but does not deliver electrical stimulation. This allows for blinding of participants to the intervention condition while maintaining the same study procedures and device usage as the active tDCS group.
  Arms: Sham tDCS

SUMMARY:
Total knee arthroplasty (TKA) is widely performed to reduce pain from advanced osteoarthritis, yet many patients experience severe postoperative pain and up to 25-44% develop chronic postsurgical pain (CPSP). Transcranial direct current stimulation (tDCS), a non-invasive neuromodulation technique, has shown promise in reducing pain and opioid use in early studies but has not been evaluated using comprehensive perioperative, home-based protocols. This study will test whether a home-based tDCS intervention delivered before and after TKA can improve acute pain management and reduce the development of CPSP.

DETAILED DESCRIPTION:
Participants will self-administer 15 tDCS sessions using a home-based device during the perioperative period. Feasibility and acceptability will be assessed through device-recorded adherence data, participant diaries completed during the intervention period, and follow-up diary entries on postoperative days 14, 30, and 90. Findings will be used to refine the protocol and inform the design of a future large-scale trial evaluating the efficacy of home-based tDCS for postoperative pain management following TKA.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. American Society of Anesthesiologists (ASA) Physical Classification Status I-III.
3. Scheduled to undergo unilateral elective primary total knee arthroplasty for advanced osteoarthritis of the knee.
4. Access to a device running iOS Version 10.0 or above, or Android Version 5.0 or above that can connect to the internet.

Exclusion Criteria:

1. History of brain surgery, central nervous system tumors, seizures (including epilepsy), stroke or intracranial implants (e.g plates, screws, deep brain stimulators)
2. Have vascular, traumatic, infectious, or metabolic lesions or diseases of the brain
3. Active diagnosis of a sleep disorder, defined as a documented diagnosis of any of the following conditions within the past 12 months, based on patient history or medical record review:

   * Insomnia disorder (e.g., difficulty initiating or maintaining sleep, early morning awakening)
   * Obstructive sleep apnea (OSA)
   * Central sleep apnea
   * Narcolepsy
   * Restless legs syndrome
   * REM sleep behavior disorder
   * Circadian rhythm sleep-wake disorders
   * Parasomnias (e.g., sleepwalking, night terrors)
4. Active diagnosis of alcohol use disorder, defined as meeting DSM-5 criteria or documented in the patient's medical record within the past 12 months.
5. Patients taking opioid medications with a daily Oral Morphine Equivalent (OME) of ≥ 80 mg
6. Current use of medications or substances known to alter cortical excitability or possess psychoactive properties (e.g., antiepileptics, benzodiazepines, antidepressants, antipsychotics, hallucinogens, dissociatives), as determined by review of the patient's medication list, chart review, and patient history. This includes prescribed medications and illicit substances used within the past 30 days.
7. Have metallic implants or objects in or on the head, including mouth (e.g. electrodes, stents, clips, pins, braces, shrapnel, jewellery (unremovable)
8. Use passive or active implanted medical devices (e.g., pacemakers, defibrillators, cochlear implants, natural implants or active body-worn medical devices (e.g., neural stimulation or medication infusion devices)
9. Have defects in the neurocranium (e.g., post-skull trepanation)
10. Have large vessel occlusions (e.g., complete blockage of the internal carotid artery or other conditions affecting brain perfusion
11. Have skin diseases of the scalp
12. Are using other brain stimulation devices concurrently
13. Are pregnant
14. Are unable to provide informed consent
15. Are unable to wear or tolerate the study device
16. Unable to speak or read English, or understand device operation instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility outcomes | Pre-op Days -5 to +90 days
  Enrollment: number of patients enrolled per week (proceed if ≥1/wk; modify protocol if 0.5-1/wk; fail to proceed if <0.5/wk) Intervention Adherence: percent of randomized participants completing all stimulation sessions (proceed if >80%; modify protocol if 50-80%; fail to proceed if <50%) Data Completeness: percent of randomized participants completing the Numeric Rating Scale pain score at end of tDCS treatment; (proceed if >85%; modify protocol if 60-85%; fail to proceed if <60%)

SECONDARY OUTCOMES:
Treatment Acceptability | Post-op 14 days
  tDCS Treatment Acceptability Questionnaire

OTHER OUTCOMES:
Pain Intensity | Post-op day 1 to 90
  Assessed using Numeric Rating Scale (NRS)
Knee-Specific Pain, Function, and Quality of Life | Post-op day 1 to 90
  Measured using the Knee Injury and Osteoarthritis Outcome Score (KOOS)
Postoperative Analgesic Medication and Opioid Use | Post-op day 1 to 90
  Self-reported and converted to oral morphine equivalents
Quality of Life Assessment | Post-op day 1 to 90
  Assessed using PROMIS-29 domain scores
Participant Blinding Success | Post-op day 1 to 90
  Evaluated using the Bang Blinding Index (BBI)
Device Related Side Effects | Post-op day 1 to 90
  Patient-Reported Side Effect Diary

CONTACTS AND LOCATIONS:
Overall Officials: Karim Ladha, MD, FRCPC, Principal Investigator — Women's College Hospital
Locations (1):
- Toronto Western Hospital (UHN), Toronto, Ontario, Canada